CLINICAL TRIAL: NCT01300741
Title: One Month Performance Comparison Between 2 Commercially Available Silicone Hydrogel Lenses
Brief Title: One Month Performance Comparison Between Two Commercially Available Silicone Hydrogel Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P-336-C-018
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Results first posted 2012-05-09 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotrafilcon B (Experimental): Lotrafilcon B commercially marketed contact lens randomly assigned to one eye, with galyfilcon A commercially marketed contact lens in the fellow eye for contralateral wear. Lenses were worn for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks in a daily wear (DW modality).
  Interventions: Device: Lotrafilcon B contact lens (AIR OPTIX® AQUA); Device: Contact lens solution (Clear Care®)
- Galyfilcon A (Active Comparator): Galyfilcon A commercially marketed contact lens randomly assigned to one eye, with lotrafilcon B commercially marketed contact lens in the fellow eye for contralateral wear. Lenses were worn for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks in a daily wear (DW modality).
  Interventions: Device: Galyfilcon A contact lens (ACUVUE® ADVANCE® Plus); Device: Contact lens solution (Clear Care®)

INTERVENTIONS:
Device: Lotrafilcon B contact lens (AIR OPTIX® AQUA) — Silicone hydrogel, single vision contact lens worn in one eye in a daily wear modality for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks.
  Other Names: AIR OPTIX® AQUA
  Arms: Lotrafilcon B
Device: Galyfilcon A contact lens (ACUVUE® ADVANCE® Plus) — Silicone hydrogel, single vision contact lens worn in one eye in a daily wear modality for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks.
  Other Names: ACUVUE® ADVANCE® Plus
  Arms: Galyfilcon A
Device: Contact lens solution (Clear Care®) — Hydrogen peroxide-based system used for cleaning, disinfection and overnight storage of the study contact lenses.
  Other Names: Clear Care®

SUMMARY:
The purpose of this study is to compare the performance of two commercially marketed contact lenses when worn for up to one month in a daily wear modality.

ELIGIBILITY:
Inclusion Criteria:

* Habitual spherical soft contact lens wearer who wears a contact lens brand with a recommended replacement schedule of 2 weeks or greater.
* Have a need for correction in both eyes and be correctable to at least 20/40 distance vision in each eye at the dispense of study lenses.
* Willing and able to wear spherical contact lenses within the available range of powers.
* Wears contact lenses at least 5 days per week and at least 10 hours per day, removing them nightly.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks prior to enrollment.
* Currently enrolled in any clinical trial.
* Any use of medications for which contact lens wear could be contraindicated, as determined by the investigator.
* Astigmatism of 1.00D or more.
* Currently wearing contact lenses in a daily disposable modality.
* Currently wearing AIR OPTIX AQUA or ACUVUE ADVANCE Plus contact lenses.
* Currently sleeping overnight in contact lenses on an occasional or extended wear basis.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 US study centers.
Groups:
- Lotrafilcon B / Galyfilcon A: Lotrafilcon B commercially marketed contact lens randomly assigned to one eye, with galyfilcon A commercially marketed contact lens in the fellow eye for contralateral wear. Lenses were worn in a daily wear (DW) modality for approximately 5 days or more per week, at least 10 hours per day, for up to 4 weeks.
Period: Overall Study
Arm/Group | Lotrafilcon B / Galyfilcon A
Started | 75
Completed | 72
Not Completed | 3
Not completed — Lens deposits | 1
Not completed — Lost to Follow-up | 1
Not completed — Discomfort | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lotrafilcon B / Galyfilcon A
Number analyzed (Participants) | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 30.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Comfort on Insertion
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Comfort on insertion was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: Analysis conducted per protocol, with exclusions due to reasons such as, major protocol deviations as determined by masked review; discontinuations; and/or missing responses
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Lotrafilcon B: Lotrafilcon B commercially marketed contact lens randomly assigned to one eye and worn for up to 4 weeks in a daily wear (DW) modality.
- Galyfilcon A: Galyfilcon A commercially marketed contact lens randomly assigned to one eye and worn for up to 4 weeks in a daily wear (DW) modality, with a replacement lens issued at 2 weeks.
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.7 (1.4) | 8.5 (1.6)

2. Primary Outcome: Comfort During the Day
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Comfort during the day was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.4 (1.5) | 8.4 (1.6)

3. Primary Outcome: Comfort at End of Day
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Comfort at end of day was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 7.8 (1.9) | 7.7 (2.0)

4. Primary Outcome: Overall Comfort
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Overall comfort was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.3 (1.7) | 8.2 (1.7)

5. Primary Outcome: Daytime Vision
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Daytime vision was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.8 (1.6) | 8.7 (1.6)

6. Primary Outcome: Low Light Vision
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Low light vision was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 68
Units on a Scale | 8.6 (1.5) | 8.5 (1.5)

7. Primary Outcome: Handling on Insertion
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Handling on insertion was graded on a 10-point scale, with 1 being difficult and 10 being easy.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.8 (1.4) | 8.6 (1.7)

8. Primary Outcome: Handling at Removal
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Handling at removal was graded on a 10-point scale, with 1 being difficult and 10 being easy.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.8 (1.5) | 8.8 (1.5)

9. Primary Outcome: Delivers a Healthy, Natural Feeling
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Delivers a healthy, natural feeling was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.6 (1.5) | 8.3 (1.9)

10. Primary Outcome: Lens Awareness
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Lens awareness was graded on a 10-point scale, with 1 being very aware and 10 being not aware.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.1 (2.1) | 7.8 (2.5)

11. Primary Outcome: Overall Satisfaction
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. Overall satisfaction was graded on a 10-point scale, with 1 being poor and 10 being excellent.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Units on a Scale | 8.4 (1.7) | 8.0 (2.0)

12. Primary Outcome: Purchase Intent
Description: As interpreted and recorded by the participant on a questionnaire as a single, retrospective evaluation of 4 weeks of wear. The participant was asked, "How likely would you be to purchase these lenses?" Purchase intent was graded on a 5-point Likert scale: Definitely would purchase, probably would purchase, may or may not purchase, probably would not purchase, definitely would not purchase. The Top-2-box response (definitely would purchase, probably would purchase) was calculated and reported as a percentage of all responses.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: Percent likely to purchase
Arm/Group | Lotrafilcon B | Galyfilcon A
Number analyzed (Participants) | 69 | 69
Percent likely to purchase | 55.1 | 56.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the trial: 16 FEB 2011 to 28 MAR 2011.
Arm/Group | Lotrafilcon B | Galyfilcon A
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.